CLINICAL TRIAL: NCT02186158
Title: Interest of Ascorbic Acid in the Management of Pneumonia in Elderly People Hospitalized.
Acronym: PNEUMO-VITA-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2013/09
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Pneumonia With Hospitalized Elderly Patient
Keywords: Pneumonia; Elderly; Ascorbic acid; Vitamin C; Hospitalized patient
MeSH Terms: conditions — Pneumonia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C (Experimental): Each patient of this group will be received a direct intravenous injection of 2,5 ml ascorbic acid twice a day (at the morning and the lunchtime) from d1 to d2 included. From d3 to d7 included, ascorbic acid's capsules produced by the University Hospital Bordeaux's central pharmacy to keep the double blind way of this study will be given at patient at the morning and at the lunchtime.
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): Each patient of this group will be received a direct intravenous injection of 2,5 ml NaCl 9% twice a day (at the morning and the lunchtime) from d1 to d2 included. From d3 to d7 included, mannitol's capsules produced by the University Hospital Bordeaux's central pharmacy will be given at patient at the morning and at the lunchtime.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C
  Arms: Vitamin C
Drug: Placebo
  Arms: Placebo

SUMMARY:
Pneumonia is the second common infection and its risk increases for elderly. In this population, it is the first cause of mortality by infections, and source of many complications. Geriatric studies had shown the high prevalence of ascorbic acid 's deficiency, especially in older hospitalized people. It is well known that vitamin C is one of the key of the immune system, it has a scavenger's role in case of aggression like sepsis. A Cochrane database published in 2013 analyzed the impact of vitamin C for preventing and treating pneumonia. Two randomized studies showed a benefit on respiratory symptoms for patients treated by vitamin C, and for one of those studies it was noted a significant reduction of mortality. The main objective of our study is first to determine the impact on respiratory symptoms of an adjuvant treatment by vitamin C for the management of pneumonia in older people hospitalized, and then evaluate its impact on functional status.

DETAILED DESCRIPTION:
This study is French non-comparative phase II clinical trial, double-blind randomized, with placebo, single-center. One group would be treated the placebo group, and another would receive an adjuvant treatment by vitamin C : 500 mg twice a day by intra-venous way from the first day to the second included, and then 500 mg twice a day by oral way from the third day to the seventh. For each patient, the study's duration is 7 days, which is the mean stay of hospitalization. During those 7 days, we will make clinical exams and blood tests at d0, d2, d4 and d7. The vitamin C blood level will be measured at d0 and d7.

ELIGIBILITY:
Inclusion Criteria:

* people aged ≥ 75 years old
* pneumonia's symptoms according to the SPILF (Société de Pathologie Infectieuse de Langue Française) :

  * cough
  * at least one respiratory sign : dyspnea, chest pain, wheezing, and local signs at the auscultation
  * at least one general sign suggesting an infection : fever, sweat, headache, sore joints, common cold
* pneumonia's symptoms developed between the admission's date in the unit care and the seventh day included

Exclusion Criteria:

* palliative care's patients
* patients with deglutition's disorders
* patients who can't be on a drip
* antibiotherapy since more one day
* other concomitant infection(s)
* patients who can't make their own transfer 15 days ago
* patients who have a NYHA score at IV 15 days ago
* patients with contraindication to a vitamin C treatment : hemochromatosis, oxalo-calcic lithiasis antecedent, G6PD deficit (Glucose 6 Phosphate Dehydrogenase), and treatment by Deferoxamine

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference in the NYHA score between d-15 and d4 after treatment initiation | 4 days after randomisation/treatment initiation
  The NYHA score d-15 would be noted by medical staff at the inclusion by calling the patient's general practitioner. The NYHA score at d4 will be noted by investigators treating the patient.

SECONDARY OUTCOMES:
The NYHA score at d2 and d7 | 2 and 7 days after randomisation/treament initiation
Dyspnea's visual analogic scale at d2, d4 and d7 | 2, 4 and 7 days after randomisation/treament initiation
Blood saturation without oxygen therapy at d2, d4 and d7 | 2, 4 and 7 days after randomisation/treament initiation
Katz's ADL (Activities Daily Living) score at d2,d4 and d7 | 2, 4 and 7 days after randomisation/treament initiation
  Katz's ADL will be calculated by medical trained students or doctors at d2, d4 and d7
Asthenia's evaluation at d2,d4 and d7 | 2, 4 and 7 days after randomisation/treament initiation
Possibility for the patient to make his or her own transfer at d2,d4 and d7 | 2, 4 and 7 days after randomisation/treament initiation
Morbidity-mortality at d2,d4 and d7 | 2, 4 and 7 days after randomisation/treament initiation
Blood inflammation parameters at d2,d4 and d7 | 2, 4 and 7 days after randomisation/treament initiation
  Leukocytes and polynuclear neutrophil 's rates, with C-reactive protein will be measured at d2, d4 and d7
Vitamin C blood level at d7 | 7 days after randomisation/treament initiation

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie LAFARGUE, MD, Principal Investigator — University Hospital Bordeaux (France); Antoine BENARD, MD, Study Chair — University Hospital Bordeaux (France)
Locations (1):
- CHU de Bordeaux, Hôpital Saint André, Bordeaux, France